CLINICAL TRIAL: NCT04273971
Title: Acute Effect of Plyometric Exercises on Musculotendinous Properties of Quadriceps and Biceps Femoral
Brief Title: Acute Effect of Plyometric Exercises on Musculotendinous Properties
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Universidade Federal de Santa Maria (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government); Federal University of Rio Grande do Sul (Other)
Responsible Party: Principal Investigator, Karine Josibel Velasques Stoelben, Principal Investigator, Universidade Federal do Pampa
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20180702141429
Record Dates: First submitted 2020-02-13; First posted 2020-02-18 (Actual); Last update posted 2020-11-05 (Actual); Status verified 2020-11

CONDITIONS: Healthy
Keywords: Adult; Lower extermity; Plyometric exercise; Muscle properties
MeSH Terms: interventions — Plyometric Exercise

STUDY DESIGN:
Intervention Model Description: Single-arm design where all participants receive treatment.
Masking Description: The statistical analyzer will be masking for the time factor.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Plyometric exercise (Experimental)
  Interventions: Other: Plyometric exercises

INTERVENTIONS:
Other: Plyometric exercises — Plyometric exercises will be composed of vertical jumps, box jumps, half squat jumps, high straight jumps, bounding jumps, drop jumps and 10-m sprint.

SUMMARY:
Preventive and rehabilitation programs include plyometric exercises to promote agility, power, and muscle activation pattern during jumping. These exercises also are known to cause a high mechanical load that increases the risk of a musculoskeletal injury. The knowledge regarding the musculoskeletal damage result from this configuration of exercise can help to elaborate safer and effective training and rehabilitation programs. In this study, the investigators will conduct a clinical trial to determine the acute effect of plyometric exercises on damage caused on different portions of quadriceps and biceps femoral's muscles and tendons of quadriceps, and biceps femoral, and its effects on mechanical properties.

DETAILED DESCRIPTION:
This is a single-arm clinical trial aiming to determine the acute effect of one session of plyometric exercises on quadriceps and biceps femoral musculotendinous properties in healthy individuals.

The sample size was determined using G*Power software considering the application of ANOVA: Repeated measures, between factors, 90% power, alpha 0.05. Data from muscle echo intensity of the rectus femoral by Muddle et al. (2019) were considered for this calculation, with an effect size 0.44. A total of 30 individuals was required for this study.

The outcomes will include the muscle and tendon quality, and mechanical properties of the tendon. The assessments will be performed at three different moments: before exercise, immediately after, and 48 hours after exercise.

The data analysis will be performed per protocol. Generalized estimating equations will be used to identify the effects of time followed by Bonferroni posthoc. When effects are found, effect sizes will be estimated. Missing data will be estimated by statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* Who practice physical activity (except jump training);
* No previous lower extremity muscle injury at least 6 months before the recruitment;
* No previous lower extremity ligament or tendon injury or surgery;
* No auditory, vestibular, visual or musculoskeletal injuries or disease that limit the execution of the exercise and assessment protocols;
* No hypertension, cardiovascular, or respiratory disease.

Exclusion Criteria:

* Body mass index greater than 30 kg/m².

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-02-20 (Actual); Primary Completion 2021-10-05 (Estimated); Study Completion 2022-03-30 (Estimated)

PRIMARY OUTCOMES:
Change from baseline of echo intensity of quadriceps and biceps femoral muscles | Baseline, immediately after exercise and up to 48 hours exercise
  Muscle echo intensity will be assessed for transversal and longitudinal ultrasonography images.
Change from baseline stiffness of patellar tendon | Baseline, immediately after exercise and up to 48 hours exercise
  Patellar tendon stiffness during 5 seconds rampa contraction protocol. Patellar tendon stiffness will be estimate from force/deformation relationship of tendon.
Change from baseline young modulus of patellar tendon | Baseline, immediately after exercise and up to 48 hours exercise
  Patellar tendon young modulus during rampa contraction protocol. Young modulus will be estimate from force/deformation relationship of tendon normalized to transverse section area of tendon.

SECONDARY OUTCOMES:
Change from baseline echo intensity of quadriceps and biceps femoral tendons | Baseline, immediately after exercise and up to 48 hours exercise
  Tendons echo intensity will be assessed for transversal and longitudinal ultrasonography images.

OTHER OUTCOMES:
Change from baseline muscle soreness of quadriceps and biceps femoral muscles | Baseline and up to 48 hours exercise
  Soreness will be measure as treashold of pain feeling while a hand-held dynamometer apply force.

CONTACTS AND LOCATIONS:
Overall Officials: Felipe P Carpes, PhD, Study Director — Universidade Federal do Pampa; Marco A Vaz, PhD, Study Chair — Federal University of Rio Grande do Sul
Locations (1):
- Karine Josibel Velasques Stoelben, Uruguaiana, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: Yes
The investigators intend to publish the results in an open-access journal, indexed at the Directory of Open Access Journals, with the copyrights transferred to the authors. Details regarding the study's design and statistical plan can be obtained consulting the trial's protocol. Data on other outcomes could be requested contacting the PI.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: The individual participant dataset will become available at a public repository up to six months after the first study publication
Access Criteria: A simple registration will grant access to study datasets. The website for these files is not defined at the time of registration.